CLINICAL TRIAL: NCT00670826
Title: Intraoperative Warming: Comparison of Performance of the Dynatherm Medical vitalHEAT Temperature Management System(vH2)With the Arizant Bair Hugger System
Brief Title: Comparison Study of Intraoperative Patient Warming Systems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dynatherm Medical Inc. (Industry)
Responsible Party: Kent Weinmeister, MD, Mayo Clinic Scottsdale
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M100 IRB07-003313; TP0010C
Record Dates: First submitted 2008-04-29; First posted 2008-05-02 (Estimated); Last update posted 2008-05-02 (Estimated); Status verified 2008-04

CONDITIONS: Orthopedic Surgery; General Anesthesia
Keywords: Patient warming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Use of the Dynatherm Medical vitalHEAT vH2 Temperature Management System to warm patients undergoing orthopedic surgical procedures with an expected duration 2-3 hours and requiring general anesthesia.
  Interventions: Device: vitalHEAT vH2 Temperature Management System
- 2 (Active Comparator): Use of the Arizant Healthcare Bair Hugger Temperature Management System & Bair Hugger Upper Body Blanket to warm patients undergoing orthopedic surgical procedures with an expected duration 2-3 hours and requiring general anesthesia.
  Interventions: Device: Arizant Healthcare Bair Hugger Temperature Management System

INTERVENTIONS:
Device: vitalHEAT vH2 Temperature Management System — The vH2 system utilizes a combination of localized heat and vacuum application to one hand & forearm; this application opens AVAs in the palm of the hand and warms the extremity thus effectively warming the blood flowing to the body's core.
  Arms: 1
Device: Arizant Healthcare Bair Hugger Temperature Management System — The Bair Hugger system is a forced air system providing convective warming via the circulation of warmed air through specially designed blanket which is placed over a portion of the body
  Arms: 2

SUMMARY:
Medications used to put people to sleep during surgical procedures also cause changes in the body's ability to control its temperature. These changes can make a person's temperature drop below normal. To minimize this drop in body temperature, different types of body warming products are used during surgery. This study is designed to compare the the temperatures of people under general anesthesia after 60 minutes of warming with each product. The study hypothesis is that the people warmed with the Dynatherm Medical vitalHEAT vH2 System will decrease less in the first 60 minutes of warming time than people warmed with the Arizant Bair Hugger System.

ELIGIBILITY:
Inclusion Criteria:

* Pts undergoing orthopedic surgical procedure with expected duration 2-3 hrs
* General anesthesia required
* ASA physical status I-III

Exclusion Criteria:

* General anesthesia plus epidural anesthesia required
* Skin abrasions/trauma to extremity selected as application site
* History of peripheral vascular disease
* History of malignant hyperthermia
* Unwilling/unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-09 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Compare esophageal temperatures after 60 minutes of warming with each system | 60 minutes of patient warming

SECONDARY OUTCOMES:
Compare esophageal temperature trends during surgical procedures | Every 15 minutes during procedure
Compare sublingual temperatures of patients in PACU | Within 10 minutes of arrival in PACU

CONTACTS AND LOCATIONS:
Overall Officials: Kent P Weinmeister, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Hospital, Phoenix, Arizona, United States